CLINICAL TRIAL: NCT00744211
Title: Proteolytic Enzyme Induction Within the Human Myocardial Interstitium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SURG-001-07F
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Results first posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Heart Disease
MeSH Terms: conditions — Heart Diseases | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vehicle (Placebo Comparator): Vehicle Group
  Interventions: Other: Vehicle
- ET-ARA 1mg/kg (Experimental): ET-ARA 1 mg/kg
  Interventions: Drug: 1mg/kg sitaxsentan sodium
- ET-ARA 2mg/kg (Experimental): ET-ARA 2 mg/kg
  Interventions: Drug: 2mg/kg sitaxsentan sodium

INTERVENTIONS:
Drug: 1mg/kg sitaxsentan sodium — 1mg/kg sitaxsentan sodium (intravenous bolus) performed immediately before separation from cardiopulmonary bypass and again at 12 hours after cardiopulmonary bypass.
  Other Names: TBC11251Na
  Arms: ET-ARA 1mg/kg
Drug: 2mg/kg sitaxsentan sodium — 2mg/kg sitaxsentan sodium (intravenous bolus) performed immediately before separation from cardiopulmonary bypass and again at 12 hours after cardiopulmonary bypass.
  Other Names: TBC11251Na
  Arms: ET-ARA 2mg/kg
Other: Vehicle — Intravenous bolus performed immediately before separation from cardiopulmonary bypass and again at 12 hours after cardiopulmonary bypass.
  Other Names: Saline
  Arms: Vehicle

SUMMARY:
A robust release of endothelin-1-1 (ET) with subsequent ETA subtype receptor (ET-AR) activation occurs in patients following cardiac surgery requiring cardiopulmonary bypass (CPB). Increased ET-AR activation has been identified in patients with poor left ventricular (LV) function (reduced ejection fraction; EF). Accordingly, this study tested the hypothesis that a selective ET-AR antagonist (ET-ARA) administered peri-operatively would favorably affect post-CPB hemodynamic profiles in patients with a pre-existing poor LVEF.

DETAILED DESCRIPTION:
Patients with a reduced LVEF were prospectively randomized, in a blinded fashion, at the time of elective coronary revascularization and/or valve replacement requiring CPB, to infusion of the highly-selective and potent ET-ARA, sitaxsentan at 1 or 2 mg/kg (IV bolus) or vehicle (saline). Infusion of the ET-ARA/vehicle was performed immediately prior to separation from CPB and again at 12 hrs post-CPB. ET and hemodynamic measurements were performed at baseline, at separation from CPB (Time 0) and at 0.5, 6, 12, 24 hrs post-CPB.

ELIGIBILITY:
Inclusion Criteria:

* >60 years of age
* Body mass index <40 kg/m2
* Left ventricular ejection fraction less than or equal to 50% documented by a pre-operative echocardiogram
* Patients undergoing coronary artery bypass (CABG), aortic and/or mitral valve replacement or combined CABG and valve procedures requiring CPB.
* If diabetic, be under proper control, (fasting glucose <350 mg/dL or recent hemoglobin A1c [HgbA1c] <9%).
* If hypertensive, be on a stable medical regimen with no significant changes over the past 30 days.
* Female of child bearing potential with a negative pregnancy test, or post-menopausal for at least 2 years
* The patient is an appropriate study candidate as determined by the Investigator on the basis of medical history and physical examination

Exclusion Criteria:

* Emergent revascularization
* Previous stroke or thrombo-embolic event in the 3 months prior to study entry
* A previous myocardial infarction within the last 7 days
* Documented coagulopathy
* Hepatic dysfunction as defined by aspartate transaminase (AST) or alanine transaminase (ALT) > 1.5 times the upper limit of normal
* Patient is pregnant or breastfeeding

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-07; Primary Completion 2011-06 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Spinale, MD PhD, Principal Investigator — Wm. Jennings Bryan Dorn VA Medical Center, Columbia, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Spinale FG, Koval CN, Deschamps AM, Stroud RE, Ikonomidis JS. Dynamic changes in matrix metalloprotienase activity within the human myocardial interstitium during myocardial arrest and reperfusion. Circulation. 2008 Sep 30;118(14 Suppl):S16-23. doi: 10.1161/CIRCULATIONAHA.108.786640. PMID 18824748
- [Result] Ford RL, Mains IM, Hilton EJ, Reeves ST, Stroud RE, Crawford FA Jr, Ikonomidis JS, Spinale FG. Endothelin-A receptor inhibition after cardiopulmonary bypass: cytokines and receptor activation. Ann Thorac Surg. 2008 Nov;86(5):1576-83. doi: 10.1016/j.athoracsur.2008.06.076. PMID 19049753
- [Result] Toole JM, Ikonomidis JS, Szeto WY, Zellner JL, Mulcahy J, Deardorff RL, Spinale FG. Selective endothelin-1 receptor type A inhibition in subjects undergoing cardiac surgery with preexisting left ventricular dysfunction: Influence on early postoperative hemodynamics. J Thorac Cardiovasc Surg. 2010 Mar;139(3):646-54. doi: 10.1016/j.jtcvs.2009.11.046. Epub 2010 Jan 13. PMID 20074751

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective randomization in a blinded fashion, at the time of elective coronary revascularization or valve replacement requiring cardiopulmonary bypass.
Groups:
- Vehicle: Saline intravenous bolus
- ET-ARA 1mg/kg: 1mg/kg sitaxsentan sodium intravenous bolus
- ET-ARA 2mg/kg: 2mg/kg sitaxsentan sodium intravenous bolus
Period: Baseline
Arm/Group | Vehicle | ET-ARA 1mg/kg | ET-ARA 2mg/kg
Started | 10 | 9 | 10
Completed | 10 | 9 | 10
Not Completed | 0 | 0 | 0
Period: 0.5 Hours After Cardiopulmonary Bypass
Arm/Group | Vehicle | ET-ARA 1mg/kg | ET-ARA 2mg/kg
Started | 10 | 9 | 10
Completed | 10 | 9 | 10
Not Completed | 0 | 0 | 0
Period: 6 Hours After Cardiopulmonary Bypass
Arm/Group | Vehicle | ET-ARA 1mg/kg | ET-ARA 2mg/kg
Started | 10 | 9 | 10
Completed | 10 | 9 | 10
Not Completed | 0 | 0 | 0
Period: 12 Hours After Cardiopulmonary Bypass
Arm/Group | Vehicle | ET-ARA 1mg/kg | ET-ARA 2mg/kg
Started | 10 | 9 | 10
Completed | 10 | 9 | 10
Not Completed | 0 | 0 | 0
Period: 24 Hours After Cardiopulmonary Bypass
Arm/Group | Vehicle | ET-ARA 1mg/kg | ET-ARA 2mg/kg
Started | 10 | 9 | 10
Completed | 10 | 9 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Vehicle: Saline, intravenous bolus
- ET-ARA 1mg/kg: 1mg/kg sitaxsentan sodium
- ET-ARA 2mg/kg: 2mg/kg sitaxsentan sodium
- Total: Total of all reporting groups
Arm/Group | Vehicle | ET-ARA 1mg/kg | ET-ARA 2mg/kg | Total
Number analyzed (Participants) | 10 | 9 | 10 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (2) | 62 (3) | 68 (3) | 66 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 3
  Male | 9 | 7 | 10 | 26
Left Ventricular Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: percent] | 35 (3) | 38 (2) | 37 (3) | 37 (2)
Plasma Endothelin [Mean (Standard Deviation); unit: fmol/mL] | 3.9 (0.4) | 3.7 (0.3) | 4.3 (0.7) | 4.0 (0.3)
Systemic vascular resistance [Mean (Standard Deviation); unit: dyne*second/centimeter˄5] | 1408 (119) | 1359 (210) | 1307 (112) | 1358 (83)
Pulmonary vascular resistance [Mean (Standard Deviation); unit: dyne*second/centimeter˄5] | 153.8 (19.9) | 213.0 (65.3) | 174.6 (28.4) | 180 (23)

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Vascular Resistance
Description: Pulmonary Vascular Resistance (d.s.cm-5)
Time Frame: Baseline, 0, 6, 12 and 24 hours post-cardiopulmonary bypass (CPB)
Measure: Mean (Standard Deviation); unit: dyne*second/centimeter˄5
Groups:
- 1mg/kg ET-ARA: 1 mg/kg ET-ARA
- 2mg/kg ET-ARA: 2 mg/kg ET-ARA
Arm/Group | Vehicle | 1mg/kg ET-ARA | 2mg/kg ET-ARA
Number analyzed (Participants) | 10 | 9 | 10
dyne*second/centimeter˄5
  Baseline | 153.8 (19.9) | 213.0 (65.3) | 174.6 (28.4)
  0 hours post-CPB | 123.5 (20.7) | 125.3 (24.8) | 175.8 (26.6)
  6 hours post-CPB | 138.7 (28.0) | 144.6 (15.2) | 132.7 (17.6)
  12 hours post-CPB | 146.8 (21.6) | 132.7 (12.7) | 136.6 (17.5)
  24 hours post-CPB | 163.3 (26.6) | 125.5 (22.3) | 138.7 (20.0)
Statistical Analysis 1: Comparison: Vehicle vs 1mg/kg ET-ARA vs 2mg/kg ET-ARA; Test type: Superiority or Other; p < 0.05, ANOVA — p<0.05; Pairwise tests of individual groups means were compared by adjusted probabilities (Bonferroni method)

2. Secondary Outcome: Plasma Endothelin-1
Description: Plasma Endothelin-1 (fmol/mL)
Time Frame: Baseline, 0, 6, 12 and 24 hours post-CPB
Measure: Mean (Standard Deviation); unit: fmol/mL
Arm/Group | Vehicle | 1mg/kg ET-ARA | 2mg/kg ET-ARA
Number analyzed (Participants) | 10 | 9 | 10
fmol/mL
  Baseline | 3.9 (0.4) | 3.7 (0.3) | 4.3 (0.7)
  0 hours post-CPB | 5.5 (0.8) | 4.7 (0.5) | 4.1 (0.5)
  6 hours post-CPB | 8.2 (1.1) | 7.2 (1.3) | 7.6 (1.2)
  12 hours post-CPB | 8.6 (1.1) | 8.8 (1.7) | 10.4 (1.6)
  24 hours post-CPB | 8.0 (1.0) | 8.3 (1.0) | 8.6 (1.4)
Statistical Analysis 1: Comparison: Vehicle vs 1mg/kg ET-ARA vs 2mg/kg ET-ARA; Test type: Superiority or Other; p = 0.001, ANOVA — Pairwise tests of individual groups means were compared by adjusted probabilities (Bonferroni method)

3. Other Pre Specified Outcome: Sitaxsentan Levels
Description: Sitaxsentan levels (microg/mL)
Time Frame: 0, 6, 12 and 24 hours post-CPB
Measure: Mean (Standard Deviation); unit: microg/mL
Arm/Group | 1mg/kg ET-ARA | 2mg/kg ET-ARA
Number analyzed (Participants) | 9 | 10
microg/mL
  0 hours post-CPB | 7.35 (0.83) | 11.78 (1.17)
  6 hours post-CPB | 0.06 (0.01) | 2.24 (2.13)
  12 hours post-CPB | 1.88 (1.26) | 8.63 (3.24)
  24 hours post-CPB | 0.06 (0.01) | 0.09 (0.01)
Statistical Analysis 1: Comparison: 1mg/kg ET-ARA vs 2mg/kg ET-ARA; Test type: Superiority or Other; p < 0.05, ANOVA

4. Other Pre Specified Outcome: Number of Other Adverse Events By Type
Description: Other (non-serious) Adverse Events (reported by arm/group)
Time Frame: up to 24-hours post-CPB
Measure: Number; unit: events
Arm/Group | Vehicle | 1mg/kg ET-ARA | 2mg/kg ET-ARA
Number analyzed (Participants) | 10 | 9 | 10
events
  Cardiovascular | 12 | 20 | 17
  Pulmonary | 3 | 4 | 8
  Neurological | 2 | 0 | 0
  Urinary | 2 | 0 | 3
  Gastrointestinal | 9 | 8 | 8
  Hepatic | 0 | 3 | 1
  Musculoskeletal | 1 | 7 | 5
  Genitourinary/Gynecological | 0 | 0 | 0
  Endocrine/Metabolic | 1 | 1 | 5
  Immunological/Allergic | 0 | 1 | 0
  Hematological/Lymphatic | 1 | 4 | 10
  Psychological/Behavioral | 3 | 4 | 7
  HEENT | 1 | 0 | 0
  Infection | 3 | 0 | 2
  Fever | 0 | 3 | 4
  Dermatological | 0 | 3 | 2
Statistical Analysis 1: Comparison: Vehicle vs 1mg/kg ET-ARA vs 2mg/kg ET-ARA; Test type: Equivalence — Chi-square tests for differences between groups; p = 0.015, Chi-squared — P-value is associated with the hematological/lymphatic adverse event

ADVERSE EVENTS:
Time Frame: Post-operative period, reported up to 30+ days post CPB
Description: Data for the Number of Participants Affected with Other Adverse Events is no longer available. Other Adverse Event Data is only available as a count of occurrences of AE's by Arm/Group.
Groups:
- ET-ARA 1mg/kg: ET - ARA 1 mg / kg
- ET-ARA 2mg/kg: ET - ARA 2 mg / kg
Arm/Group | Vehicle | ET-ARA 1mg/kg | ET-ARA 2mg/kg
Serious Adverse Events (participants affected / at risk) | 6/10 | 6/9 | 6/10
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=10) | ET-ARA 1mg/kg (N=9) | ET-ARA 2mg/kg (N=10)
Death (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) — Following adjudication, all 3 deaths were determined to be unrelated to ET-ARA treatment.
Thrombo-embolic event (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 3 (3) — When all SAE's were considered as a composite, there were no significant differences between treatment groups (Chi-square 1.59; p=0.452).
Pulmonary/infection (Infections and infestations) | 4 (4) | 0 (0) | 2 (2) — When all SAE's were considered as a composite, there were no significant differences between treatment groups (Chi-square 1.59; p=0.452).
Gastrointestinal (ischemic bowel) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — When all SAE's were considered as a composite, there were no significant differences between treatment groups (Chi-square 1.59; p=0.452).

LIMITATIONS AND CAVEATS:
Small sample size, which in turn can result in a disproportionate number of patients with greater pre-operative risk profiles randomized to one treatment group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes